CLINICAL TRIAL: NCT00246545
Title: Effect Evaluation of Early Exercise Training After Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: fase I
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
The aim of the study is to evaluate the effect of early onset of exercise training (ET) after myocardial infarction (MI) in a randomized controlled trial. Usual care is to wait 4-6 weeks after onset of MI, and our hypotheses are that early ET will prevent a fall in VO2peak and contribute to better quality of life.

DETAILED DESCRIPTION:
Exercise training is well documented as effective treatment for myocardial infarction(MI) patients. However, the long time effect of early onset is more unclear, and it is needed to provide knowledge about to which extend early onset of ET contribute to reduce risk factors, increase oxygen consumption and influence on quality of life.

A RCT is conducted, 60 persons with recently MI is invited to participate. The subjects participating is hospitalised in St. Olavs Hospital. The participants are randomised to either a training group or a control group. The training group will be offered hospital out-patient group exercise training of moderate intensity twice a week for four weeks. The training is leaded by a physiotherapist. The control group will wait four weeks before both groups continue ET twice a week for 12 weeks (high intensity training).

ELIGIBILITY:
Inclusion Criteria:

* Myocardiac infarction, 2 weeks ago
* over 18 years
* able to participate i exercise groups

Exclusion Criteria:

* unstable angina
* heart failure
* failure to reach a maximal pretest
* drug abuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen consumption

SECONDARY OUTCOMES:
quality of life
change in risk factors (smoking habits, physical activity)

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Støylen, Dr.med, Study Director — NTNU, St.Olavs hospital; Ingerlise Aamot, PT, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Aamot IL, Moholdt T, Amundsen BH, Solberg HS, Morkved S, Stoylen A. Onset of exercise training 14 days after uncomplicated myocardial infarction: a randomized controlled trial. Eur J Cardiovasc Prev Rehabil. 2010 Aug;17(4):387-92. doi: 10.1097/HJR.0b013e328333edf9. PMID 19940774